## INFORMED CONSENT FORM

This study you participated in is a scientific research and the name of the research is "The Effect of Creative Drama Education on Attitudes Regarding Violence Against Women: A Randomized Controlled Trial" for Alcohol-Substance Addicted Male Patients. Addiction is a chronic, recurrent, needing state that creates physical and psychological distress when it is not taken. If the addictive substance is taken in high doses or not taken at all, physiological and psychological symptoms occur in individuals. As a result of these symptoms, unhappiness, conflict, aggression and violent behavior between people cause the emergence and increase. Women can be most often affected by these aggressive behaviors. In this study, a training will be applied to you when it is your turn. For the research, you are asked to participate in the trainings completely and to fill out the attached forms completely. In addition, you will need to allocate an average of 10-15 minutes to fill out the forms. Your participation in the research will contribute to the literature. The number of people to be included in this study is everyone who was in the service during the time period of the study. There are no risks or benefits for you in this research. If there are any developments during the investigation that may be of interest to you, you or your legal representative will be notified immediately. To get additional information about the research or for any problems, unwanted effects or other ailments related to the study, you can either address "Bolu İzzet Baysal Mental Health and Diseases Hospital" or call 0374-375-2525 no.lu. You can apply to Hümeyra Hançer Tok.

You will not be paid for your participation in this research and you will not be charged any fees for all examinations, examinations, tests and medical care services within the scope of this research.

Taking part in this research is entirely at your will. You may refuse to take part in the research or you may leave the research at any stage; this will not lead to any punishment or obstruction of your benefits. The researcher may remove you from the research for reasons such as not fulfilling the requirements of the treatment scheme, disrupting the study program or increasing the effectiveness of the treatment, etc. within your knowledge or against your will. The results of the research will be used for scientific purposes; If you withdraw from the study or are removed by the researcher, the medical data about you may also be used for scientific purposes if necessary.

All of your medical and identification information will be kept confidential and your identity information will not be provided even if the research is published, but the researchers, pollers, ethics committees and official authorities may access your medical information when necessary. You can also access your own medical information when you want.

## **Approval to Participate in the Study:**

I read and listened verbally to the information above that should have been given to the volunteer before the research was started. I have asked all the questions that come to my mind to the researcher, and I have understood in detail all the explanations made to me, both written and oral. I was given enough time to decide if I wanted to participate in the study. Under these circumstances, I authorize the research coordinator to review, transfer and process my medical information and voluntarily accept the invitation to participate in this research without any coercion or pressure.

I will be provided with a signed copy of this form.

| Volunteer's, | The researcher who made the statements, |
|---|---|
| Name-Surname: | Name-Surname: Hümeyra Hançer Tok |
| Address: | Position:Nurse |
| TelFax: | Address: Bolu Mental Health and Diseases Hospital |
| | TelFax:544-600-4410 |
| Date and Signature: | Date and Signature: |
| A parent or guardian for those under custody or guardianship, | The organization officer/interview witness who witnessed the |
| | consent process from the beginning to the end, |
| Name-Surname: | Name-Surname: |
| Address: | Task: |
| TelFax: | Address: |
| | TelFax: |
| Date and Signature: | |
| | Date and Signature: |

<sup>\*</sup> This sample form has been prepared by giving the minimum information that should be included in the form to give an idea to the researchers, and additions should be made when necessary. It can be used when requested by obtaining it from the secretariat of the Ethics Committee or from the Faculty of Medicine website and making the necessary arrangements on it (e.g. this paragraph, the dotted parts and parentheses in the text should be removed and arranged appropriately). The declaration and signature of the volunteer must be in the form of a continuation of the information text; it should definitely not be on separate pages. Date of update 28.11.2013